CLINICAL TRIAL: NCT02401321
Title: A Pilot Feasibility Study: Taking Care of Her
Brief Title: Taking Care of Her Program in Patients With Stage III or IV Ovarian Cancer and Spouse Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 9306; NCI-2015-00325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9306 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Caregiver; Stage IIIA Ovarian Cancer; Stage IIIB Ovarian Cancer; Stage IIIC Ovarian Cancer; Stage IV Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive care (Taking Care of Her program) (Experimental): Patients and spouse caregivers complete the Taking Care of Her Program comprising 5 telephone-delivered intervention sessions over 45-60 minutes every 2 weeks. The intervention sessions are designed to provide training for spouse caregivers and patients to better manage the impact and emotional toll of recently diagnosed ovarian cancer, including its impact on their interpersonal communication and support about the cancer.
  Interventions: Behavioral: Telephone-Based Intervention; Other: Caregiver-Assisted Training; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Behavioral: Telephone-Based Intervention — Complete Taking Care of Her program
Other: Caregiver-Assisted Training — Complete Taking Care of Her program
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot clinical trial studies the Taking Care of Her program in patients with stage III or IV ovarian cancer and spouse caregivers. This counseling program may equip the spouse caregiver with skills to support and nurture the patient through initial diagnosis and treatment. It may also help patients and spouse caregivers improve communication and coping skills.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the feasibility of the study protocol, including recruitment and retention.

II. Assess the short-term impact of the intervention on standardized measures of behavioral-emotional adjustment of spouse caregivers and diagnosed women on depressed mood, anxiety, quality of marital communication, perceived spousal support, and spouse caregivers' skills and self-confidence to manage the emotional toll of the illness on themselves and the ill partner.

OUTLINE:

Patients and spouse caregivers complete the Taking Care of Her Program comprising 5 telephone-delivered intervention sessions over 45-60 minutes every 2 weeks. The intervention sessions are designed to provide training for spouse caregivers and patients to better manage the impact and emotional toll of recently diagnosed ovarian cancer, including its impact on their interpersonal communication and support about the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Spouses of women with diagnosed within the past 8 months with stage III or IV ovarian cancer will be eligible to participate, as will the diagnosed wife/partner
* Spouses and patients must be married or cohabiting and in intimate relationship for at least 6 months
* Have English as one of their languages of choice (they can be multilingual)
* Have access to a telephone
* Have not been diagnosed with a prior cancer within the recent 5 years, except basal or squamous cell skin carcinoma
* Both heterosexual and same sex couples will be eligible

Exclusion Criteria:

* Women diagnosed with stage IV ovarian cancer and who are hospice eligible
* Spouses/partners could not participate if the patient refused participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-06-23 (Actual)

PRIMARY OUTCOMES:
Recruitment | Up to 1 year
  To test the feasibility of the study protocol, including recruitment, a detailed spreadsheet will be used to track the relative success of different recruitment channels. The channel through which every eligible patient is recruited will be tracked: self-referral, provider referral, or passive letter referral. The enrollment method that yielded the most accruals will be computed. The proportion of enrolled study participants that came from each channel used for the referral will be reported.
Retention | Up to 1 year
  The retention rate for each enrolled study participant will be reported and a detailed log of reasons for attrition will be retained.
Changes in depressed mood assessed by the Center for Epidemiologic Studies- Depression and Patient Health Questionniare-9 | Baseline to 3 months
  The short-term impact of the intervention on standardized measures of behavioral-emotional adjustment of spouse caregivers and diagnosed women on depressed mood will be assessed. If the distribution of the data are approximately normal, parametric statistics will be used to test the impact of the intervention on post-intervention scores using paired t-tests, 2-tailed, p = .05.
Changes in anxiety assessed by the State-Trait Anxiety Inventory | Baseline to 3 months
  The short-term impact of the intervention on standardized measures of behavioral-emotional adjustment of spouse caregivers and diagnosed women on anxiety will be assessed. If the distribution of the data are approximately normal, parametric statistics will be used to test the impact of the intervention on post-intervention scores using paired t-tests, 2-tailed, p = .05.
Changes in quality of marital communication assessed by the Mutuality & Interpersonal Sensitivity Scale, Total and subscales: Open Communication & Expressing Sad Feelings | Baseline to 3 months
  The short-term impact of the intervention on standardized measures of behavioral-emotional adjustment of spouse caregivers and diagnosed women on the quality of marital communication will be assessed. If the distribution of the data are approximately normal, parametric statistics will be used to test the impact of the intervention on post-intervention scores using paired t-tests, 2-tailed, p = .05.
Changes in perceived spousal support assessed by the What My Partner Does for Me Questionnaire | Baseline to 3 months
  The short-term impact of the intervention on standardized measures of behavioral-emotional adjustment of spouse caregivers and diagnosed women on perceived spousal support will be assessed. If the distribution of the data are approximately normal, parametric statistics will be used to test the impact of the intervention on post-intervention scores using paired t-tests, 2-tailed, p = .05.
Changes in spouse caregivers' skills and self-confidence to manage the emotional toll of the illness on themselves and ill partner assessed by the Cancer Self-Efficacy Scale: Total and subscales Self- and Wife/Partner-focused | Baseline to 3 months
  The short-term impact of the intervention on standardized measures of behavioral-emotional adjustment of spouse caregivers and diagnosed women on spouse caregivers' skills and self-confidence to manage the emotional toll of the illness on themselves and ill partner will be assessed. If the distribution of the data are approximately normal, parametric statistics will be used to test the impact of the intervention on post-intervention scores using paired t-tests, 2-tailed, p = .05.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Lewis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States